CLINICAL TRIAL: NCT04953728
Title: TEA for Study Participants With IBS-C Optimization of TEA Modalities for Treatment of IBS-C: A Phase 1 25 Study Participant Clinical Trial of Transcutaneous Electrical Acustimulation (TEA) in Study Participants With IBS-C
Brief Title: Optimization of Transcutaneous Electrical Acustimulation (TEA) Modalities for Treatment of IBS-C
Acronym: TEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Transtimulation Research, Inc (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Jiande Chen, Professor of Internal Medicine, Medical School, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00189911; 1UG3NS115108-01A1 (NIH)
Record Dates: First submitted 2021-06-28; First posted 2021-07-08 (Actual); Results first posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-01

CONDITIONS: IBS; Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Masking Description: All participants will receive all treatments including sham comparator in a randomized order. Participants will not be informed of which treatment they will be receiving or the treatment order to which they are assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Subjects with IBS-C (Experimental): All participants will receive all treatment options. Each participant will receive all of the following treatments; 100 Hz ST36, 100 Hz PC6, 25 Hz ST36, 25 Hz PC6, as well as the sham comparator. Each administration will be performed on different dates, between 1 and 3 weeks apart.
  Interventions: Device: Transcutaneous Electrical Acustimulation (TEA)

INTERVENTIONS:
Device: Transcutaneous Electrical Acustimulation (TEA) — Each participant will undergo 5 sessions total at two different frequencies (25 Hz and 100Hz) with electrodes placed at two different locations (wrist and knee) and a placebo session.

SUMMARY:
This study aims to determine the most effective treatment with Transcutaneous Electrical Acustimulation (TEA) for Irritable Bowel Syndrome with Constipation (IBS-C) by comparing efficacy between 5 separate sessions. The rectum pressure as measured by a device called a barostat will be compared between visits. Each session will be testing a different combination of frequency and body position of the electrodes. Electrodes placed at either the wrist or knee will be stimulated at either 25 Hz or 100 Hz.

DETAILED DESCRIPTION:
This study aims to discern whether acute, single-session Transcutaneous Electrical Acustimulation (TEA) at acupuncture points ST36 or PC6 will relieve abdominal pain induced by rectal distension in patients with IBS-C. Each study participant will have 5 research visits at the Michigan Medicine GI physiology lab. During these visits, participants will undergo a procedure similar to Anal Rectal Manometry (ARM) performed by the GI physiology lab staff. TEA is similar to this procedure as it uses the barostat device and is performed by the GI physiology lab staff. This device has a rubber catheter that will be inserted 5-15 cm into the rectum of the study participant. Then the GI physiology staff will inflate the catheter. Study participants will then be asked when they can sense the catheter. Then the GI physiology staff will continue to inflate the catheter and the study participants feel discomfort (described as the 'urge to defecate'). Then the study participant will be asked to pass the balloon (like they would pass a bowel movement).

The difference between ARM procedure and the study procedure is that there will be stimulation of acupuncture point ST36 which is below the knee cap or stimulation of acupuncture point PC6 which is just above the wrist. For this study, this mild electrical stimulation will occur simultaneously with the barostat procedure.

At each visit there will be stimulation of only one of the points at either 100Hz or 25Hz. These are the potential combinations: ST36 100Hz, ST36-25Hz, PC6-100Hz, PC6-25Hz, Sham-TEA.

The frequency and position combination (or sham visit) is randomly assigned. The randomization determines the order in which the study participant moves through the study. Every study participant will, in the end, complete one visit at each frequency and a sham visit. The study participant will also complete surveys at the appointment.

The TEA device is classified by the FDA as a non-significant risk device.

ELIGIBILITY:
Inclusion Criteria:

* Willing to comply with all study procedures and be available for the duration of the study
* Diagnosed with IBS-C satisfying Rome IV criteria
* Have symptoms present for at least the last 3 months
* Have abdominal pain that is not adequately relieved at the time of screening and the time of randomization
* Has a Visual Analog Scale (VAS) pain score of >3 (on 0-10 score)

Exclusion Criteria:

* Have an unrelated active disorder which may involve abdominal pain, such as inflammatory bowel disease, diabetes, unstable thyroid disease
* Have history of abdominal surgery (other than cholecystectomy or appendectomy)
* Are taking anticoagulants or antispasmodic, antidiarrheal, or opioids or other pain relief medications and cannot stop these medications for three consecutive days before each study visit
* Are pregnant or lactating; women of child bearing potential complete a pregnancy test at each visit
* Have known allergic reactions to components of the ECG electrodes
* Received treatment with an investigational drug or other intervention within 6 months of the date of consent
* Anything that, in the opinion of the investigator, would place the study participant at increased risk or preclude the study participant's full compliance with or completion of the study
* Are unable to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiande Chen, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data will not be shared. However, the study protocol and the study results will be shared

REFERENCES:
- [Background] Ma D, Han JS, Diao QH, Deng GF, Ping XJ, Jin WJ, Wu LZ, Cui CL, Li XD. Transcutaneous electrical acupoint stimulation for the treatment of withdrawal syndrome in heroin addicts. Pain Med. 2015 May;16(5):839-48. doi: 10.1111/pme.12738. PMID 25989154
- [Background] Jiang Y, Liu J, Liu J, Han J, Wang X, Cui C. Cerebral blood flow-based evidence for mechanisms of low- versus high-frequency transcutaneous electric acupoint stimulation analgesia: a perfusion fMRI study in humans. Neuroscience. 2014 May 30;268:180-93. doi: 10.1016/j.neuroscience.2014.03.019. Epub 2014 Mar 20. PMID 24657460
- [Background] Qu F, Wang FF, Wu Y, Zhou J, Robinson N, Hardiman PJ, Pan JX, He YJ, Zhu YH, Wang HZ, Ye XQ, He KL, Cui L, Zhao HL, Ye YH. Transcutaneous Electrical Acupoint Stimulation Improves the Outcomes of In Vitro Fertilization: A Prospective, Randomized and Controlled Study. Explore (NY). 2017 Sep-Oct;13(5):306-312. doi: 10.1016/j.explore.2017.06.004. Epub 2017 Jun 30. PMID 28915981
- [Background] Yu Y, Wei R, Liu Z, Xu J, Xu C, Chen JDZ. Ameliorating Effects of Transcutaneous Electrical Acustimulation Combined With Deep Breathing Training on Refractory Gastroesophageal Reflux Disease Mediated via the Autonomic Pathway. Neuromodulation. 2019 Aug;22(6):751-757. doi: 10.1111/ner.13021. Epub 2019 Jul 26. PMID 31347247
- [Background] Zhang B, Xu F, Hu P, Zhang M, Tong K, Ma G, Xu Y, Zhu L, Chen JDZ. Needleless Transcutaneous Electrical Acustimulation: A Pilot Study Evaluating Improvement in Post-Operative Recovery. Am J Gastroenterol. 2018 Jul;113(7):1026-1035. doi: 10.1038/s41395-018-0156-y. Epub 2018 Jun 21. PMID 29925916

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was opened in May 2021, and the first participant was consented July 1, 2021. Recruitment closed in September 2022.
Period: Overall Study
Arm/Group | Subjects With IBS-C
Started (Started means randomized to treatment but not, necessarily, receiving any treatment.) | 23
ST36 100 HZ | 20
ST36 25 HZ | 20
PC6 100 HZ | 20
PC6 25 HZ | 19
Sham 25 HZ | 22
Completed (Completed means all participants for whom all treatments were administered.) | 19
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Subjects With IBS-C: All participants will receive all treatment options. Each participant will receive all of the following treatments; 100 Hz ST36, 100 Hz PC6, 25 Hz ST36, 25 Hz PC6, as well as the sham comparator. Each administration will be performed on different dates, between 1 to 3 weeks apart.
  Transcutaneous Electrical Acustimulation (TEA): Each participant will undergo 5 sessions total at two different frequencies (25 Hz and 100Hz) with electrodes placed at two different locations (wrist and knee) and a placebo session.
Arm/Group | Subjects With IBS-C
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.26 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 17
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23
Pressure of Maximum Tolerance [Mean (Standard Deviation); unit: mmHg] — Pressure of Maximum Tolerance of the Rectum as Measured by a Barostat Device Pre TEA Administration Population: Only data from participants who were administered all treatments (19 participants) was analyzed to ensure pre- and post-comparisons by individual. Where data is presented for only 18 participants, 1 participant at baseline did not reach a maximum tolerance even at the maximum-offered pressure.
  mmHg
    Average baseline maximum tolerance of subjects pre ST36 100Hz: number analyzed (Participants) | 18
    Average baseline maximum tolerance of subjects pre ST36 100Hz | 47.22 (9.74)
    Average baseline maximum tolerance of subjects pre ST36 25Hz: number analyzed (Participants) | 19
    Average baseline maximum tolerance of subjects pre ST36 25Hz | 45.53 (10.12)
    Average baseline maximum tolerance of subjects pre PC6 100Hz: number analyzed (Participants) | 18
    Average baseline maximum tolerance of subjects pre PC6 100Hz | 47.22 (9.27)
    Average baseline maximum tolerance of subjects pre PC6 25Hz: number analyzed (Participants) | 18
    Average baseline maximum tolerance of subjects pre PC6 25Hz | 49.17 (10.18)
    Average baseline maximum tolerance of subjects pre sham: number analyzed (Participants) | 18
    Average baseline maximum tolerance of subjects pre sham | 46.39 (10.26)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pressure of Maximum Tolerance in mmHg of the Rectum as Measured by a Barostat Device When Compared to Pre-TEA Administration.
Description: The barostat device will measure the pressure changes in the rectum during controlled distension, as measured in mmHg. The study participant's maximum tolerance of distention will be compared to tolerance pre and post TEA, as well as comparing each administration to the other modalities and the sham. Higher numbers represent a higher degree of tolerance.
  Each participant came in for 1 treatment in 1 session on each of 5 separate days. The sequence of treatments each participant received over the course of their sessions was randomized per participant. In each session, a new baseline was established, because individuals' pain/discomfort may have changed over time between sessions. Each change value listed below represents the mean of the differences between each participant's tolerance with stimulation and that participant's baseline for that day.
Time Frame: Baseline data collected up to 12 minutes; participants rested for 15 minutes; 15 minutes of treatment was administered, then rectum was distended again with treatment for up to 12 minutes. Between each of 5 sessions, participants had 1-3 weeks off.
Population: Data was analyzed only for participants who received all 5 treatments to avoid the compounding impact of day-to-day variations. In the case of PC6 100 HZ, post-treatment value is missing for 1 participant.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Subjects With IBS-C
Number analyzed (Participants) | 19
mmHg
  Change in avg max tolerance per person: value at ST36 100Hz minus value at that day's baseline | 0.79 (1.80)
  Change in avg max tolerance per person: value at ST36 25Hz minus value at that day's baseline | 1.32 (2.26)
  Change in avg max tolerance per person: value at PC6 100Hz minus value at that day's baseline: number analyzed (Participants) | 18
  Change in avg max tolerance per person: value at PC6 100Hz minus value at that day's baseline | -4.44 (2.45)
  Change in avg max tolerance per person: value at PC6 25Hz minus value at that day's baseline | -4.21 (3.40)
  Change in avg max tolerance per person: value at sham minus value at that day's baseline | 1.84 (1.03)
Statistical Analysis 1: Comparison: Subjects With IBS-C; Change in maximum tolerance in mmHg of the rectum during ST36 100Hz when compared to baseline; Test type: Superiority; p = 0.77306724, t-test, 2 sided
Statistical Analysis 2: Comparison: Subjects With IBS-C; Change in maximum tolerance in mmHg of the rectum during ST36 25Hz when compared to baseline; Test type: Superiority; p = 0.24, t-test, 2 sided
Statistical Analysis 3: Comparison: Subjects With IBS-C; Change in maximum tolerance in mmHg of the rectum during PC6 100Hz when compared to baseline; Test type: Superiority; p = 0.45, t-test, 2 sided
Statistical Analysis 4: Comparison: Subjects With IBS-C; Change in maximum tolerance in mmHg of the rectum during PC6 25Hz when compared to baseline; Test type: Superiority; p = 0.13, t-test, 2 sided
Statistical Analysis 5: Comparison: Subjects With IBS-C; Change in maximum tolerance in mmHg of the rectum during Sham when compared to baseline; Test type: Superiority; p = 0.14, t-test, 2 sided

2. Primary Outcome: Change in Pressure of Maximum Tolerance in mmHg of the Rectum as Measured by a Barostat Device When Compared to Other Modalities.
Description: The barostat device measured the pressure changes in the rectum during controlled distension, as measured in mmHg. The study participant's maximum tolerance of distention was compared to tolerance pre and post TEA, as well as comparing each administration to the other modalities and the sham for that person. Higher numbers represent a higher degree of tolerance. Scores were compared between modalities of body position (ST36 or PC6), frequency (100 Hz or 25 Hz), and sham.
  Each participant came in for 1 treatment in 1 session on each of 5 separate days. The sequence of treatments each participant received over the course of their sessions was randomized per participant. Analysis is shown as a difference in treatment-induced change between different treatment modalities rather than a comparison between the average maximums under 1 treatment or another for the group as a whole.
Time Frame: After 15 minutes of treatment, rectum was distended incrementally with treatment for up to 12 minutes. Because between sessions, participants had 1-3 weeks off, the maximum time between 1 maximum-tolerated distension and another was 12 weeks.
Population: For each of the rows of data below, data from 19 participants at one treatment are compared with data from either 19 or 18 participants in the other treatment.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Subjects With IBS-C
Number analyzed (Participants) | 19
mmHg
  Change in avg max tolerance per person: value at ST36 100Hz minus value at ST36 25Hz | -0.53 (2.03)
  Change in avg max tolerance per person: value at ST36 100Hz minus value at PC6 100Hz | -1.66 (1.04)
  Change in avg max tolerance per person: value at ST36 100Hz minus value at PC6 25Hz | 5.00 (2.60)
  Change in avg max tolerance per person: value at ST36 100Hz minus value at sham | -1.05 (1.42)
  Change in avg max tolerance per person: value at ST36 25Hz minus value at PC6 100Hz | -1.13 (1.26)
  Change in avg max tolerance per person: value at ST36 25Hz minus value at PC6 25Hz | 5.53 (2.83)
  Change in avg max tolerance per person: value at ST36 25Hz minus value at sham | -0.53 (1.64)
  Change in avg max tolerance per person: value at PC6 100Hz minus value at PC6 25Hz | 6.66 (1.84)
  Change in avg max tolerance per person: value at PC6 100Hz minus value at sham | 0.61 (0.65)
  Change in avg max tolerance per person: value at PC6 25Hz minus value at sham | -6.05 (2.22)
Statistical Analysis 1: Comparison: Subjects With IBS-C; Change in average maximum tolerance of ST36 100Hz when compared to ST36 25Hz; Test type: Superiority; p = 0.81019363, t-test, 2 sided
Statistical Analysis 2: Comparison: Subjects With IBS-C; Change in average maximum tolerance of ST36 100Hz when compared to PC6 100Hz; Test type: Superiority; p = 0.18, t-test, 2 sided
Statistical Analysis 3: Comparison: Subjects With IBS-C; Change in average maximum tolerance of ST36 100Hz when compared to PC6 25Hz; Test type: Superiority; p = 0.21, t-test, 2 sided
Statistical Analysis 4: Comparison: Subjects With IBS-C; Change in average maximum tolerance of ST36 100Hz when compared to Sham; Test type: Superiority; p = 0.58, t-test, 2 sided
Statistical Analysis 5: Comparison: Subjects With IBS-C; Change in average maximum tolerance of ST36 25Hz when compared to PC6 100Hz; Test type: Superiority; p = 0.18, t-test, 2 sided
Statistical Analysis 6: Comparison: Subjects With IBS-C; Change in average maximum tolerance of ST36 25Hz when compared to PC6 25Hz; Test type: Superiority; p = 0.18, t-test, 2 sided
Statistical Analysis 7: Comparison: Subjects With IBS-C; Change in average maximum tolerance of ST36 25Hz when compared to sham; Test type: Superiority; p = 0.78, t-test, 2 sided
Statistical Analysis 8: Comparison: Subjects With IBS-C; Change in average maximum tolerance of PC6 100Hz when compared to PC6 25Hz; Test type: Superiority; p = 0.89, t-test, 2 sided
Statistical Analysis 9: Comparison: Subjects With IBS-C; Change in average maximum tolerance of PC6 100Hz when compared to sham; Test type: Superiority; p = 0.05, t-test, 2 sided
Statistical Analysis 10: Comparison: Subjects With IBS-C; Change in average maximum tolerance of PC6 25Hz when compared to sham; Test type: Superiority; p = 0.07, t-test, 2 sided

3. Secondary Outcome: Change in Pain as Measured by Visual Analog Scale (VAS) Surveys When Compared to Pre-TEA Administration.
Description: VAS surveys, a pain scale from 0 (lowest) to 10 (highest), were taken to assess efficacy of treatment on a 10-point scale. The minimum possible score was 0 and the maximum possible score was 80, if a participant experienced 10/10 pain. These scores were collected at 15 through 50 mmHg of distension at 5-mmHg intervals during baseline and compared to the scores collected at the same intervals during treatment on the same day. Data below show values post stimulation minus pre stimulation.
  Each participant came in for 1 treatment in 1 session on each of 5 separate days. Sequence of treatments each participant received over the course of their sessions was randomized per participant. In each session, a new baseline was established, because individuals' pain/discomfort may have changed over time between sessions. Analysis is shown as a single arm rather than a cross-over because the averages below are calculated from the change in each participant's pain compared only to their own pain.
Time Frame: Up to 8 mins between 15 and 50 mmHg during baseline. After deflating balloon, 15 mins of treatment and resumption of distention (up to 30 mins later), more surveys were taken during treatment increasing distensions up to 8 mins between 15 and 50 mmHg.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Subjects With IBS-C
Number analyzed (Participants) | 19
score on a scale
  ST36 100Hz | -7.74 (1.82)
  ST36 25Hz | -0.94 (2.84)
  PC6 100Hz | -4.19 (2.41)
  PC6 25Hz | -2.23 (1.87)
  Sham | -3.74 (1.77)
Statistical Analysis 1: Comparison: Subjects With IBS-C; ST36 100Hz: Difference of VAS sums between 15 and 50 mmHg between pre and post stimulation; Test type: Superiority; p = 0.00046998, t-test, 2 sided
Statistical Analysis 2: Comparison: Subjects With IBS-C; ST36 25Hz: Difference of VAS sums between 15 and 50 mmHg between pre and post stimulation; Test type: Superiority; p = 0.74369428, t-test, 2 sided
Statistical Analysis 3: Comparison: Subjects With IBS-C; PC6 100Hz: Difference of VAS sums between 15 and 50 mmHg between pre and post stimulation; Test type: Superiority; p = 0.09854383, t-test, 2 sided
Statistical Analysis 4: Comparison: Subjects With IBS-C; PC6 25Hz: Difference of VAS sums between 15 and 50 mmHg between pre and post stimulation; Test type: Superiority; p = 0.24872746, t-test, 2 sided
Statistical Analysis 5: Comparison: Subjects With IBS-C; Sham: Difference of VAS sums between 15 and 50 mmHg between pre and post stimulation; Test type: Superiority; p = 0.04828889, t-test, 2 sided

4. Secondary Outcome: Change in Individual's Pain as Measured by Visual Analog Scale (VAS) Surveys at Max Distension During 1 Treatment Compared to Their Own Pain During a Different Treatment.
Description: VAS surveys, a pain scale from 0 (lowest) to 10 (highest), were taken to assess efficacy of treatment on a 10-point scale. The minimum possible score is 0 and the maximum possible score is 80, if a participant experienced 10/10 pain. These scores, collected at maximum distension during treatment, were compared between modalities of body position (ST36 or PC6), frequency (100 Hz or 25 Hz), and sham for each individual.
  Each participant came in for 1 treatment in 1 session on each of 5 separate days. The sequence of treatments each participant received over the course of their sessions was randomized per participant. Analysis is shown as a difference in treatment-induced change between different treatment modalities rather than a comparison between the average pain scores under 1 treatment or another for the group as a whole.
Time Frame: Surveys taking less than 1 minute were taken at maximum-tolerated distension during treatment. Because between sessions, participants had 1-3 weeks off, the maximum time between 1 survey and another was 12 weeks.
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Subjects With IBS-C
Number analyzed (Participants) | 19
score on a scale
  Change in VAS per person: value at ST36 100Hz minus value at ST36 25Hz | -6.80 (2.33)
  Change in VAS per person: value at ST36 100Hz minus value at PC6 100Hz | -3.55 (2.11)
  Change in VAS per person: value at ST36 100Hz minus value at PC6 25Hz | -5.51 (1.84)
  Change in VAS per person: value at ST36 100Hz minus value at Sham | -3.99 (1.79)
  Change in VAS per person: value at ST36 25Hz minus value at PC6 100Hz | 3.25 (2.62)
  Change in VAS per person: value at ST36 25Hz minus value at PC6 25Hz | 1.29 (2.35)
  Change in VAS per person: value at ST36 25Hz minus value at Sham | 2.80 (2.30)
  Change in VAS per person: value at PC6 100Hz minus value at PC6 25Hz | -1.96 (2.14)
  Change in VAS per person: value at PC6 100Hz minus value at Sham | -0.45 (2.09)
  Change in VAS per person: value at PC6 25Hz minus value at Sham | 1.52 (1.82)
Statistical Analysis 1: Comparison: Subjects With IBS-C; ST36 100Hz compared to ST36 25Hz; Test type: Superiority; p = 0.02, t-test, 1 sided
Statistical Analysis 2: Comparison: Subjects With IBS-C; ST36 100Hz compared to PC6 100Hz; Test type: Superiority; p = 0.11, t-test, 1 sided
Statistical Analysis 3: Comparison: Subjects With IBS-C; ST36 100Hz compared to PC6 25Hz; Test type: Superiority; p = 0.01, t-test, 1 sided
Statistical Analysis 4: Comparison: Subjects With IBS-C; ST36 100Hz compared to Sham; Test type: Superiority; p = 0.04, t-test, 1 sided
Statistical Analysis 5: Comparison: Subjects With IBS-C; ST36 25Hz compared to PC6 100Hz; Test type: Superiority; p = 0.11, t-test, 1 sided
Statistical Analysis 6: Comparison: Subjects With IBS-C; ST36 25Hz compared to PC6 25Hz; Test type: Superiority; p = 0.23, t-test, 1 sided
Statistical Analysis 7: Comparison: Subjects With IBS-C; ST36 25Hz compared to Sham; Test type: Superiority; p = 0.17, t-test, 1 sided
Statistical Analysis 8: Comparison: Subjects With IBS-C; PC6 100Hz compared to PC6 25Hz; Test type: Superiority; p = 0.15, t-test, 1 sided
Statistical Analysis 9: Comparison: Subjects With IBS-C; PC6 100Hz compared to Sham; Test type: Superiority; p = 0.43, t-test, 1 sided
Statistical Analysis 10: Comparison: Subjects With IBS-C; PC6 25Hz compared to Sham; Test type: Superiority; p = 0.19, t-test, 1 sided

5. Secondary Outcome: Change in Maximum Volume in mL of the Rectum as Measured by a Barostat Device When Compared to Pre-TEA Administration.
Description: The barostat device will measure the volume changes in the rectum during controlled distension, as measured in milliliters. The study participant's maximum volume will be compared to tolerance pre and post TEA. A higher number corresponds to a higher maximum volume.
  Each participant came in for 1 treatment in 1 session on each of 5 separate days. The sequence of treatments each participant received over the course of their sessions was randomized per participant. In each session, a new baseline was established, because individuals' maximum volume may have changed over time between sessions. Each change value listed below represents the mean of the differences between each participant's maximum volume with stimulation and that participant's baseline for that day. Analysis is shown as a single arm rather than a cross-over because the averages below are calculated from the change in each participant's maximum volume compared only to their own maximum volume.
Time Frame: as for outcome 1
Population: Data from participants who did not reach a maximum tolerance at a preset maximum distension pressure of 60 mmHg were not analyzed. For some participants, the barostat was unable to provide complete data to allow analysis.
Measure: Mean (Standard Error); unit: mL
Arm/Group | Subjects With IBS-C
Number analyzed (Participants) | 19
mL
  Change in max vol per participant in mL of the rectum during ST36 100Hz minus max vol at baseline: number analyzed (Participants) | 18
  Change in max vol per participant in mL of the rectum during ST36 100Hz minus max vol at baseline | -2.31 (13.59)
  Change in max vol per participant in mL of the rectum during ST36 25Hz minus max vol at baseline: number analyzed (Participants) | 15
  Change in max vol per participant in mL of the rectum during ST36 25Hz minus max vol at baseline | 14.08 (8.74)
  Change in max vol per participant in mL of the rectum during PC6 100Hz minus max vol at baseline: number analyzed (Participants) | 15
  Change in max vol per participant in mL of the rectum during PC6 100Hz minus max vol at baseline | 11.83 (8.10)
  Change in max vol per participant in mL of the rectum during PC6 25Hz minus max vol at baseline: number analyzed (Participants) | 16
  Change in max vol per participant in mL of the rectum during PC6 25Hz minus max vol at baseline | -1.56 (10.01)
  Change in max vol per participant in mL of the rectum during sham minus max vol at baseline: number analyzed (Participants) | 17
  Change in max vol per participant in mL of the rectum during sham minus max vol at baseline | 13.48 (8.75)
Statistical Analysis 1: Comparison: Subjects With IBS-C; Change in maximum volume in mL of the rectum during ST36 100Hz when compared to baseline; Test type: Superiority; p = 0.87, t-test, 2 sided
Statistical Analysis 2: Comparison: Subjects With IBS-C; Change in maximum volume in mL of the rectum during ST36 25Hz when compared to baseline; Test type: Superiority; p = 0.13, t-test, 2 sided
Statistical Analysis 3: Comparison: Subjects With IBS-C; Change in maximum volume in mL of the rectum during PC6 100Hz when compared to baseline; Test type: Superiority; p = 0.17, t-test, 2 sided
Statistical Analysis 4: Comparison: Subjects With IBS-C; Change in maximum volume in mL of the rectum during PC6 25Hz when compared to baseline; Test type: Superiority; p = 0.88, t-test, 2 sided
Statistical Analysis 5: Comparison: Subjects With IBS-C; Change in maximum volume in mL of the rectum during sham when compared to baseline; Test type: Superiority; p = 0.14, t-test, 2 sided

6. Secondary Outcome: Change in Pressure of First Sensation of the Rectum as Measured by a Barostat Device When Compared to Pre-TEA Administration.
Description: The barostat device measured the pressure changes in the rectum during controlled distension, as measured in mmHg. Values below show the pressure at which each participant experienced first sensation of the rectum during stimulation minus the pressure at which each participant experienced first sensation at baseline.
  Each participant came in for 1 treatment in 1 session on each of 5 separate days. The sequence of treatments each participant received over the course of their sessions was randomized per participant. In each session, a new baseline was established, because individuals' pressure may have changed over time between sessions. Analysis is shown as a single arm rather than a cross-over because the averages below are calculated from the change in each participant's pressure compared only to their own pressure.
Time Frame: as for outcome 1
Population: In the case of PC6 100 HZ, post-treatment value is missing for 1 participant.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Subjects With IBS-C
Number analyzed (Participants) | 19
mmHg
  ST36 100Hz | 5.79 (1.88)
  ST36 25Hz | 0.26 (1.18)
  PC6 100Hz: number analyzed (Participants) | 18
  PC6 100Hz | 1.87 (0.97)
  PC6 25Hz | 6.05 (1.82)
  Sham | 2.63 (1.29)
Statistical Analysis 1: Comparison: Subjects With IBS-C; Change in first sensation in mmHg of the rectum during ST36 100Hz when compared to baseline; Test type: Superiority; p = 0.007, t-test, 2 sided
Statistical Analysis 2: Comparison: Subjects With IBS-C; Change in first sensation in mmHg of the rectum during ST36 25Hz when compared to baseline; Test type: Superiority; p = 0.83, t-test, 2 sided
Statistical Analysis 3: Comparison: Subjects With IBS-C; Change in first sensation in mmHg of the rectum during PC6 100Hz when compared to baseline; Test type: Superiority; p = 0.87, t-test, 2 sided
Statistical Analysis 4: Comparison: Subjects With IBS-C; Change in first sensation in mmHg of the rectum during PC6 25Hz when compared to baseline; Test type: Superiority; p = 0.004, t-test, 2 sided
Statistical Analysis 5: Comparison: Subjects With IBS-C; Change in first sensation in mmHg of the rectum during sham when compared to baseline; Test type: Superiority; p = 0.056, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from first visit of the study to one month after the last visit of the study, a maximum of 16 weeks.
Description: Data in this module is presented under each treatment. The treatments do not represent separate arms.
Groups:
- ST36 100 HZ: Administration of 100 HZ to acupressure point ST36
- ST36 25 HZ: Administration of 25 HZ to acupressure point ST36
- PC6 100 HZ: Administration of 100 HZ to acupressure point PC6
- PC6 25 HZ: Administration of 25 HZ to acupressure point PC6
- Sham 25 HZ: Administration of 25 HZ to sham acupressure point
Arm/Group | ST36 100 HZ | ST36 25 HZ | PC6 100 HZ | PC6 25 HZ | Sham 25 HZ
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/19 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/19 | 0/22
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 1/20 | 0/19 | 2/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ST36 100 HZ (N=20) | ST36 25 HZ (N=20) | PC6 100 HZ (N=20) | PC6 25 HZ (N=19) | Sham 25 HZ (N=22)
Hematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1) — Noticed 7 days after the previous study visit where sham stimulation was administered.
Belching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1) — belching occurred after completion of the first distension and prior to sham stimulation
Hematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 — Noticed upon removal of balloon after PC6-100Hz stimulation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT04953728/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT04953728/ICF_002.pdf